CLINICAL TRIAL: NCT07363798
Title: Association of Nutrition and T Cell Immune Activity With Disease Progression in Nontuberculous Mycobacterial Pulmonary Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Deog Kyeom Kim, Clinical Professor, Department of Pulmonary and Critical Care Medicine, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Other Study IDs: BRMH 20-2025-65
Record Dates: First submitted 2025-12-26; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Disease; Nontuberculous Mycobacterial Lung Disease
Keywords: Nontuberculous mycobacterial pulmonary disease; Bronchoalveolar lavage; T cell exhaustion; Disease progression; Nutritional status
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NTM-PD cohort: This cohort includes adults (≥18 years) with confirmed or suspected nontuberculous mycobacterial pulmonary disease (NTM-PD) in whom active pulmonary tuberculosis has been excluded and who are undergoing bronchoscopy as part of routine clinical care. Participants receive standard-of-care evaluation and management according to established NTM clinical guidelines. There are no experimental interventions assigned in this study. Residual bronchoalveolar lavage fluid remaining after clinically indicated testing is used for immunologic analyses, including flow cytometric assessment of inhibitory and exhausted T-cell subsets. Clinical data, nutritional status, imaging findings, and laboratory results are collected prospectively, and participants are followed longitudinally to assess time to initiation of antimicrobial treatment due to clinical disease progression and other clinically relevant outcomes.

SUMMARY:
Nontuberculous mycobacterial pulmonary disease (NTM-PD) is a chronic lung infection caused by environmental mycobacteria. The clinical course of NTM-PD varies widely among patients. Some individuals remain stable for long periods without treatment, while others experience worsening lung disease that requires antibiotic therapy or may lead to death. Currently available clinical tools are limited in their ability to predict which patients will experience disease progression.

This observational study aims to better understand how the body's immune response and nutritional status are related to disease progression in adults with confirmed or suspected NTM-PD. In particular, the study focuses on T cells, a type of immune cell that plays an important role in controlling mycobacterial infections. Prior research suggests that impaired T-cell function may contribute to disease progression in NTM-PD, but most studies have relied on blood samples rather than immune cells from the lung, where the infection occurs.

In this study, immune cells obtained from bronchoalveolar lavage fluid during clinically indicated bronchoscopy will be analyzed to assess inhibitory and exhausted T-cell profiles in the lung. In addition, systemic T-cell function will be evaluated using the mitogen response from the QuantiFERON-TB Gold Plus blood test. Nutritional status and body composition will also be assessed, as poor nutrition is known to affect immune function and disease outcomes.

Participants will be followed over time as part of routine clinical care. The primary outcome of the study is the time from enrollment to the initiation of antibiotic treatment due to clinical disease progression. Secondary outcomes include identifying immune predictors of treatment initiation, examining the relationship between nutritional status and immune activity, evaluating changes in body composition and immune markers with disease progression, and determining whether immune and nutritional measures improve prediction of mortality beyond established clinical risk scores.

By integrating lung immune profiling, blood-based immune testing, nutritional assessment, and clinical data, this study seeks to improve risk stratification in NTM-PD. The results may help identify patients at higher risk for disease progression and poor outcomes, support more personalized monitoring strategies, and inform future studies targeting immune and nutritional pathways in NTM-PD.

DETAILED DESCRIPTION:
Nontuberculous mycobacterial pulmonary disease (NTM-PD) is a chronic and heterogeneous infectious lung disease caused by a variety of environmental mycobacteria, including Mycobacterium avium complex (MAC), Mycobacterium abscessus subspecies, Mycobacterium kansasii, and other rapidly or slowly growing species. Despite increasing global prevalence, the clinical course of NTM-PD remains highly variable. Some patients experience long-term stability without treatment, whereas others develop progressive lung destruction, recurrent exacerbations, treatment failure, or death. This heterogeneity highlights limitations in current prognostic tools and underscores the need for biologically informed risk stratification.

The BACES score (Body mass index <18.5 kg/m², Age ≥65 years, Cavitary disease, Elevated erythrocyte sedimentation rate, and male Sex) is a validated clinical scoring system for mortality prediction in NTM-PD. While clinically practical, BACES relies exclusively on demographic, nutritional, inflammatory, and radiographic variables and does not incorporate direct measures of host immune function. Increasing evidence suggests that host immune dysregulation-particularly impairment of adaptive T-cell-mediated immunity-plays a central role in disease progression and may explain outcome differences among patients with similar clinical features.

Recent translational studies using lung tissue, spatial transcriptomics, and peripheral blood immunophenotyping have demonstrated a characteristic immune imbalance in NTM-PD. These studies consistently show hyperactivation of innate immune pathways (e.g., macrophage and monocyte inflammatory signaling) alongside functional suppression of T-cell-mediated adaptive immunity. This T-cell dysfunction is characterized by reduced antigen-specific interferon-gamma (IFN-γ) production, decreased co-stimulatory signaling (such as CD28 downregulation), and increased expression of inhibitory immune checkpoint receptors, including programmed death-1 (PD-1) and T-cell immunoglobulin and mucin-domain containing-3 (TIM-3). Additionally, CD39-expressing T cells-associated with adenosine-mediated immunosuppression and terminal exhaustion-have been implicated in chronic infectious and inflammatory states.

Importantly, increased frequencies of PD-1-positive or TIM-3-positive CD4+ T cells have been associated with higher mycobacterial burden, cavitary disease, low body mass index, and adverse clinical outcomes in NTM-PD. These inhibitory and exhausted T-cell phenotypes appear to reflect chronic antigenic stimulation and impaired immune control of infection. However, most prior studies have relied on peripheral blood samples, which may not accurately represent the immune microenvironment within the lung, the primary site of disease activity.

Bronchoalveolar lavage (BAL) fluid provides direct access to immune cells within affected lung segments and offers a unique opportunity to characterize local pulmonary immune responses. BAL-derived T-cell immunophenotyping may therefore yield more clinically relevant insights into disease pathogenesis and progression than blood-based analyses alone. Nonetheless, systematic evaluation of inhibitory and exhausted T-cell subsets in BAL fluid and their association with clinically meaningful outcomes in NTM-PD remains limited.

In parallel, systemic T-cell functional capacity may influence disease trajectory. The QuantiFERON-TB Gold Plus assay includes a mitogen control that measures nonspecific T-cell interferon-gamma production. The Mitogen minus Nil value reflects overall T-cell immune reserve independent of antigen specificity. Low mitogen responses have been associated with immune suppression, severe infection, prolonged hospitalization, and increased mortality in other clinical contexts. Despite its widespread clinical use, the prognostic relevance of the QuantiFERON mitogen response has not been systematically evaluated in NTM-PD.

Nutritional status represents another key modulator of immune function. Low body mass index, reduced muscle mass, and diminished fat reserves are well-established risk factors for NTM-PD development and progression. Nutritional deficiency is also known to impair T-cell metabolism, proliferation, cytokine production, and memory formation. Thus, nutritional status may interact with immune dysfunction to influence disease outcomes. Integrating nutritional, immunologic, and clinical data may therefore enable a more comprehensive understanding of NTM-PD progression.

Study Objectives

This prospective observational study is designed to investigate whether bronchoalveolar lavage-derived inhibitory and exhausted T-cell profiles and systemic T-cell functional capacity, assessed by the QuantiFERON mitogen response, are associated with time to initiation of antimicrobial treatment due to clinical disease progression in adults with confirmed or suspected NTM-PD. Furthermore, the study aims to determine whether incorporating these immune and nutritional parameters into established clinical risk models, including the BACES score, improves prognostic discrimination for clinically meaningful outcomes, including treatment initiation and all-cause mortality.

Study Design and Population

This is a single-center, prospective observational cohort study enrolling adults aged 18 years or older with confirmed or suspected NTM-PD in whom active pulmonary tuberculosis has been excluded. Eligible participants are those undergoing bronchoscopy as part of routine clinical evaluation or disease monitoring according to established NTM management guidelines. No additional invasive procedures are performed solely for research purposes.

Patients with active tuberculosis, current malignancy requiring treatment, solid organ or stem cell transplantation, systemic immunosuppressive therapy, autoimmune disease, recent acute lower respiratory tract infection, or pregnancy are excluded to minimize confounding effects on immune function.

Sample Collection and Immunologic Assessment

Bronchoalveolar lavage is performed according to standard clinical protocols. After completion of all clinically indicated diagnostic testing, residual BAL fluid is processed for flow cytometric analysis. BAL cells are filtered, washed, and stained with a multicolor antibody panel designed to characterize T-cell lineage, activation status, regulatory features, and inhibitory and exhausted phenotypes.

Key immunologic parameters include:

* Frequencies of CD4+ and CD8+ T cells expressing PD-1, TIM-3, and CD39
* Co-expression patterns of inhibitory immune checkpoint receptors
* Regulatory T-cell populations defined by CD25^high and CD127^low expression
* Co-stimulatory marker expression (CD28)
* T-cell subset differentiation states relevant to chronic antigen exposure and immune exhaustion

Peripheral blood laboratory data are obtained from routine clinical testing. QuantiFERON-TB Gold Plus results are collected, with particular emphasis on the Mitogen minus Nil value as a measure of global T-cell functional capacity.

Nutritional and Radiographic Assessment

Nutritional status is assessed using anthropometric measurements (body mass index, waist circumference), the Mini Nutritional Assessment questionnaire, and body composition metrics derived from clinically indicated chest computed tomography. Quantitative measurements include skeletal muscle area and subcutaneous and visceral fat compartments at standardized anatomical levels using validated image analysis software.

Radiographic disease severity is evaluated using chest CT-based scoring systems that account for the extent of nodules, bronchiectasis, consolidation, and cavitary lesions. Disease phenotype (e.g., nodular bronchiectatic or fibrocavitary form) is recorded.

Follow-up and Outcomes

Participants are followed longitudinally according to routine clinical practice, typically at 3- to 6-month intervals. Follow-up evaluations include sputum mycobacterial cultures, radiographic imaging, and clinical assessments.

The primary outcome is time to initiation of antimicrobial treatment due to clinical disease progression, defined as the interval from study enrollment to the start of guideline-based therapy, as determined by the treating physician based on worsening respiratory symptoms, microbiologic findings, and/or radiographic deterioration requiring treatment.

Secondary outcomes include:

* Immune predictors of treatment initiation, including bronchoalveolar lavage-derived inhibitory and exhausted T-cell profiles and systemic T-cell functional capacity assessed by the QuantiFERON mitogen response
* Associations between nutritional status and T-cell immune activity
* Within-participant changes in body composition and T-cell immune activity between baseline and the time of disease progression requiring treatment
* Incremental prognostic value of immune and nutritional parameters beyond the BACES score for predicting all-cause mortality

Statistical Analysis

Associations between immune parameters, nutritional variables, and clinical outcomes are evaluated using appropriate univariate and multivariable statistical methods. Time-to-event analyses are performed using Kaplan-Meier methods and Cox proportional hazards models, with time to initiation of treatment due to disease progression as the primary time-to-event outcome. Logistic regression or Cox regression models are used, as appropriate, to identify independent immune and nutritional predictors of treatment initiation.

To assess prognostic performance for mortality, models incorporating BAL-derived immune variables, QuantiFERON mitogen responses, and nutritional parameters are compared with clinical models based on the BACES score alone. Discrimination and reclassification performance are evaluated using measures such as the area under the receiver operating characteristic curve (AUROC), concordance index, and reclassification metrics where appropriate.

Significance

By integrating local pulmonary immune profiling, systemic T-cell functional assessment, nutritional evaluation, and established clinical risk scores, this study seeks to advance biologically informed risk stratification in NTM-PD. The findings may help identify patients at higher risk for treatment-requiring disease progression and mortality, support personalized monitoring strategies, and provide a foundation for future interventional studies targeting immune and nutritional pathways in NTM-PD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Confirmed or suspected nontuberculous mycobacterial pulmonary disease
* Active pulmonary tuberculosis excluded by standard microbiologic testing
* Undergoing bronchoscopy as part of routine clinical evaluation or disease monitoring
* Able and willing to provide written informed consent

Exclusion Criteria:

* Active pulmonary tuberculosis confirmed by microbiologic testing
* Positive latent tuberculosis infection test
* Current active malignancy requiring treatment
* History of solid organ transplantation or hematopoietic stem cell transplantation
* Use of systemic immunosuppressive medications
* Diagnosis of autoimmune disease
* Use of biologic agents or planned initiation of biologic therapy
* Acute lower respiratory tract infection requiring treatment within 4 weeks prior to bronchoscopy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from adults with confirmed or suspected nontuberculous mycobacterial pulmonary disease who are scheduled to undergo bronchoscopy as part of routine clinical evaluation or disease monitoring according to established NTM management guidelines. The study population consists of patients receiving standard-of-care clinical assessment and follow-up, without any additional procedures performed solely for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of treatment due to disease progression in nontuberculous mycobacterial pulmonary disease | From enrollment to initiation of nontuberculous mycobacterial treatment, up to 24 months
  Time to treatment initiation is defined as the duration from study enrollment to the start of antimicrobial therapy for nontuberculous mycobacterial pulmonary disease due to clinical disease progression. Treatment initiation is determined by the treating physician based on standard clinical practice and guideline-based criteria, including worsening respiratory symptoms, microbiologic findings, and/or radiographic deterioration indicating progression requiring treatment. This primary outcome is used to evaluate the association between time to treatment initiation and immune predictors, including bronchoalveolar lavage-derived inhibitory and exhausted T-cell profiles and systemic T-cell functional capacity, assessed by the QuantiFERON mitogen response, along with other clinical factors.

SECONDARY OUTCOMES:
Proportion of regulatory T cells in bronchoalveolar lavage fluid (BAL) at baseline | Baseline
  Regulatory T cells (Tregs) in BAL fluid are measured by flow cytometry on samples collected at baseline. The outcome is defined as the percentage of CD4⁺ T cells that express regulatory markers (CD3⁺, CD4⁺, CD25^hi, CD127^low) in the baseline BAL sample. This immune cell frequency serves as one of the baseline immune parameters in the study.
Proportion of exhausted T cells in BAL fluid at baseline | Baseline
  Exhausted T cells in BAL fluid are measured by flow cytometry at baseline. These are T cells exhibiting an "exhausted" phenotype, characterized by the expression of inhibitory receptors such as PD-1, TIM-3, or CD39. The outcome is the percentage of T cells in the BAL sample that display this exhausted phenotype (CD3⁺, CD4⁺/CD8⁺, PD-1⁺, TIM-3⁺, CD39⁺) at baseline.
QuantiFERON-TB Gold Plus mitogen response at baseline (IU/mL) | Baseline
  The QuantiFERON-TB Gold Plus assay is used to assess systemic T-cell functional capacity at baseline. The outcome is the interferon-gamma concentration (Mitogen minus Nil value, reported in IU/mL) from the mitogen-stimulated tube of the QuantiFERON assay. This value reflects the overall ability of the participant's T cells to produce IFN-γ in response to a non-specific stimulus (mitogen) at baseline.
Body Mass Index (BMI) at baseline (kg/m²) | Baseline
  BMI is calculated as weight in kilograms divided by height in meters squared (kg/m²), measured at baseline. It serves as an anthropometric indicator of the participant's nutritional status. The baseline BMI is documented for each participant as part of the nutritional assessment.
Mini Nutritional Assessment (MNA) score at baseline | Baseline
  The MNA is a validated nutrition screening tool that provides a score (ranging, for example, from 0 to 14) reflecting the participant's nutritional status. Each participant's MNA is administered at baseline, and the total score is recorded. This baseline MNA score represents the nutritional status of the participant at study entry.
Pectoralis muscle area (PMA) at baseline (cm²) | Baseline
  The cross-sectional area of the pectoralis muscles is measured on a chest CT scan at baseline. Specifically, the measurement is taken on a single axial CT image at the level just below the aortic arch, and the area is reported in square centimeters (cm²). This baseline PMA provides an indicator of skeletal muscle mass (a marker of body composition and nutritional status) at the start of the study.
Visceral fat area (VFA) at baseline (cm²) | Baseline
  Visceral fat area is measured on a CT image at baseline to quantify central adiposity. The measurement is taken on an axial CT slice at the level of the T12 vertebra, and the area of visceral adipose tissue is reported in square centimeters (cm²). This baseline VFA is recorded as a body composition parameter related to nutritional status.
Subcutaneous fat area (SFA) at baseline (cm²) | Baseline
  Subcutaneous fat area is measured on a CT image at baseline to assess peripheral adipose tissue mass. The measurement is taken on an axial CT slice at the level of the T12 vertebra, and the area of subcutaneous fat is reported in square centimeters (cm²). This baseline SFA provides another body composition metric reflecting nutritional reserves.
Change in BAL Fluid Regulatory T-Cell Proportion from Baseline to Disease Progression | At time of disease progression requiring treatment (within up to 24 months).
  The change in the proportion of regulatory T cells in BAL fluid from baseline to the time of disease progression requiring treatment. This is expressed as the percentage at progression minus the percentage at baseline of BAL T cells that are regulatory T cells. A change in this value indicates how the immunoregulatory T cell population in the lungs has shifted by the time the disease progresses.
Change in BAL Fluid Exhausted T-Cell Proportion from Baseline to Disease Progression | At time of disease progression requiring treatment (within up to 24 months)
  The change in the proportion of exhausted T cells in BAL fluid between baseline and the time of disease progression requiring treatment. This is expressed as the percentage at progression minus the percentage at baseline of BAL T cells that are exhausted T cells. A change in this value indicates how the exhausted T cell population in the lungs has shifted by the time the disease progresses.
Change in Pectoralis Muscle Area (PMA) from Baseline to Disease Progression Description | At time of disease progression requiring treatment (within up to 24 months)
  The change in PMA on chest CT, measured in square centimeters (cm²), from baseline to the time of disease progression requiring treatment. The PMA at the time of progression is compared to the baseline area, and the change is calculated as the ratio of the area at progression to the area at baseline (PMA at progression / PMA at baseline). A ratio less than 1 indicates loss of muscle mass between enrollment and the point of disease progression.
Change in Visceral Fat Area on CT at T12 Level from Baseline to Disease Progression | At time of disease progression requiring treatment (within up to 24 months)
  The change in visceral fat area (cm²) on CT at the T12 level from baseline to the time of disease progression requiring treatment. The visceral fat area at the time of progression is compared to the baseline value, and the change is calculated as the ratio of the visceral fat area at progression to that at baseline (area at progression / area at baseline). A ratio less than 1 indicates an decrease in visceral adipose tissue by the time the disease has progressed to the point of requiring therapy.
Change in Subcutaneous Fat Area on CT at T12 Level from Baseline to Disease Progression | At time of disease progression requiring treatment (within up to 24 months)
  The change in subcutaneous fat area (cm²) on CT at the T12 level from baseline to the time of disease progression requiring treatment. The subcutaneous fat area at the time of progression is compared to the baseline value, and the change is calculated as the ratio of the subcutaneous fat area at progression to that at baseline (area at progression / area at baseline). A ratio less than 1 indicates an decrease in subcutaneous adipose tissue by the time the disease has progressed to the point of requiring therapy.
All-Cause Mortality within 24 Months (Comparison of BACES vs Immune-Augmented Score) | From enrollment through 24 months of follow-up
  All-cause mortality is defined as death from any cause within 24 months of enrollment. The percentage of participants who experience all-cause mortality by 24 months will be determined. Mortality outcomes using a combined risk score (the BACES clinical score plus T-cell immune activity measures) will be compared with mortality outcomes using the BACES score alone to evaluate the incremental prognostic value of adding immune parameters. Specifically, this comparison will assess whether participants who have the same BACES score (baseline clinical risk) show different 24-month survival probabilities when an immune marker-based score (incorporating BAL Treg cell percentage, BAL exhausted T-cell percentage, and QuantiFERON mitogen response) is included. An improvement in risk stratification or discrimination with the combined score would indicate that the immune parameters provide additional prognostic information for mortality beyond the established BACES score.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Dongjak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. The study includes sensitive clinical, immunologic, and imaging data derived from bronchoalveolar lavage samples and other patient-specific assessments, and no formal data-sharing infrastructure or governance plan has been established at the time of trial registration. However, de-identified individual participant data that underlie the results reported in peer-reviewed publications may be made available after publication upon reasonable request to the corresponding author, subject to appropriate data use agreements, institutional approval, and compliance with applicable ethical and privacy regulations.

REFERENCES:
- [Result] Molwitz I, Ozga AK, Gerdes L, Ungerer A, Kohler D, Ristow I, Leiderer M, Adam G, Yamamura J. Prediction of abdominal CT body composition parameters by thoracic measurements as a new approach to detect sarcopenia in a COVID-19 cohort. Sci Rep. 2022 Apr 19;12(1):6443. doi: 10.1038/s41598-022-10266-0. PMID 35440794
- [Result] Bunk SAO, Ipema J, Sidorenkov G, Bennink E, Vliegenthart R, de Jong PA, Pompe E, Charbonnier JP, Luijk BHD, Aerts J, Groen HJM, Mohamed Hoesein FAA. The relationship of fat and muscle measurements with emphysema and bronchial wall thickening in smokers. ERJ Open Res. 2024 Mar 4;10(2):00749-2023. doi: 10.1183/23120541.00749-2023. eCollection 2024 Mar. PMID 38444665
- [Result] Diaz AA, Zhou L, Young TP, McDonald ML, Harmouche R, Ross JC, San Jose Estepar R, Wouters EF, Coxson HO, MacNee W, Rennard S, Maltais F, Kinney GL, Hokanson JE, Washko GR; ECLIPSE investigators. Chest CT measures of muscle and adipose tissue in COPD: gender-based differences in content and in relationships with blood biomarkers. Acad Radiol. 2014 Oct;21(10):1255-61. doi: 10.1016/j.acra.2014.05.013. Epub 2014 Aug 1. PMID 25088837
- [Result] Kahnert K, Jorres RA, Kauczor HU, Biederer J, Jobst B, Alter P, Biertz F, Mertsch P, Lucke T, Lutter JI, Trudzinski FC, Behr J, Bals R, Watz H, Vogelmeier CF, Welte T; COSYCONET Study-Group; Names of participating study nurses. Relationship between clinical and radiological signs of bronchiectasis in COPD patients: Results from COSYCONET. Respir Med. 2020 Oct;172:106117. doi: 10.1016/j.rmed.2020.106117. Epub 2020 Aug 22. PMID 32891937
- [Result] Kim HJ, Kwak N, Hong H, Kang N, Im Y, Jhun BW, Yim JJ. BACES Score for Predicting Mortality in Nontuberculous Mycobacterial Pulmonary Disease. Am J Respir Crit Care Med. 2021 Jan 15;203(2):230-236. doi: 10.1164/rccm.202004-1418OC. PMID 32721164
- [Result] Daley CL, Iaccarino JM, Lange C, Cambau E, Wallace RJ Jr, Andrejak C, Bottger EC, Brozek J, Griffith DE, Guglielmetti L, Huitt GA, Knight SL, Leitman P, Marras TK, Olivier KN, Santin M, Stout JE, Tortoli E, van Ingen J, Wagner D, Winthrop KL. Treatment of nontuberculous mycobacterial pulmonary disease: an official ATS/ERS/ESCMID/IDSA clinical practice guideline. Eur Respir J. 2020 Jul 7;56(1):2000535. doi: 10.1183/13993003.00535-2020. Print 2020 Jul. PMID 32636299
- [Result] Hyung K, Kim SA, Kim JY, Kwak N, Yim JJ. Rates and Risk Factors of Progression in Patients With Nontuberculous Mycobacterial Pulmonary Disease: Secondary Analysis of a Prospective Cohort Study. Chest. 2024 Sep;166(3):452-460. doi: 10.1016/j.chest.2024.03.024. Epub 2024 Mar 16. PMID 38499238
- [Result] Lindestam Arlehamn CS, Benson B, Kuan R, Dill-McFarland KA, Peterson GJ, Paul S, Nguyen FK, Gilman RH, Saito M, Taplitz R, Arentz M, Goss CH, Aitken ML, Horne DJ, Shah JA, Sette A, Hawn TR. T-cell deficiency and hyperinflammatory monocyte responses associate with Mycobacterium avium complex lung disease. Front Immunol. 2022 Oct 3;13:1016038. doi: 10.3389/fimmu.2022.1016038. eCollection 2022. PMID 36263044
- [Result] Koh J, Kim S, Kim JY, Yim JJ, Kwak N. Immunologic features of nontuberculous mycobacterial pulmonary disease based on spatially resolved whole transcriptomics. BMC Pulm Med. 2024 Aug 13;24(1):392. doi: 10.1186/s12890-024-03207-2. PMID 39138424
- [Result] Raynor JL, Chi H. Nutrients: Signal 4 in T cell immunity. J Exp Med. 2024 Mar 4;221(3):e20221839. doi: 10.1084/jem.20221839. Epub 2024 Feb 27. PMID 38411744
- [Result] Wang Q, Wu H. T Cells in Adipose Tissue: Critical Players in Immunometabolism. Front Immunol. 2018 Oct 30;9:2509. doi: 10.3389/fimmu.2018.02509. eCollection 2018. PMID 30459770
- [Result] Kim SJ, Yoon SH, Choi SM, Lee J, Lee CH, Han SK, Yim JJ. Characteristics associated with progression in patients with of nontuberculous mycobacterial lung disease : a prospective cohort study. BMC Pulm Med. 2017 Jan 5;17(1):5. doi: 10.1186/s12890-016-0349-3. PMID 28056937
- [Result] Yamazaki Y, Kubo K, Takamizawa A, Yamamoto H, Honda T, Sone S. Markers indicating deterioration of pulmonary Mycobacterium avium-intracellulare infection. Am J Respir Crit Care Med. 1999 Dec;160(6):1851-5. doi: 10.1164/ajrccm.160.6.9902019. PMID 10588596
- [Result] Kim SJ, Park J, Lee H, Lee YJ, Park JS, Cho YJ, Yoon HI, Lee CT, Lee JH. Risk factors for deterioration of nodular bronchiectatic Mycobacterium avium complex lung disease. Int J Tuberc Lung Dis. 2014 Jun;18(6):730-6. doi: 10.5588/ijtld.13.0792. PMID 24903946
- [Result] Kartalija M, Ovrutsky AR, Bryan CL, Pott GB, Fantuzzi G, Thomas J, Strand MJ, Bai X, Ramamoorthy P, Rothman MS, Nagabhushanam V, McDermott M, Levin AR, Frazer-Abel A, Giclas PC, Korner J, Iseman MD, Shapiro L, Chan ED. Patients with nontuberculous mycobacterial lung disease exhibit unique body and immune phenotypes. Am J Respir Crit Care Med. 2013 Jan 15;187(2):197-205. doi: 10.1164/rccm.201206-1035OC. Epub 2012 Nov 9. PMID 23144328
- [Result] Kim RD, Greenberg DE, Ehrmantraut ME, Guide SV, Ding L, Shea Y, Brown MR, Chernick M, Steagall WK, Glasgow CG, Lin J, Jolley C, Sorbara L, Raffeld M, Hill S, Avila N, Sachdev V, Barnhart LA, Anderson VL, Claypool R, Hilligoss DM, Garofalo M, Fitzgerald A, Anaya-O'Brien S, Darnell D, DeCastro R, Menning HM, Ricklefs SM, Porcella SF, Olivier KN, Moss J, Holland SM. Pulmonary nontuberculous mycobacterial disease: prospective study of a distinct preexisting syndrome. Am J Respir Crit Care Med. 2008 Nov 15;178(10):1066-74. doi: 10.1164/rccm.200805-686OC. Epub 2008 Aug 14. PMID 18703788
- [Result] Takayama Y, Kitajima T, Honda N, Sakane N, Yumen Y, Fukui M, Nagai N. Nutritional status in female patients with nontuberculous mycobacterial lung disease and its association with disease severity. BMC Pulm Med. 2022 Aug 15;22(1):315. doi: 10.1186/s12890-022-02109-5. PMID 35971083